CLINICAL TRIAL: NCT02308579
Title: Prevalence of Chronic Cerebrospinal Venous Insufficiency in Patients With Multiple Sclerosis and Other Neurological Diseases. An Ultrasound, Blinded, Case-Controlled, Centralized Reading Assessment
Brief Title: Centralized Reading Assessment of Chronic CerebroSpinal Venous Insufficiency (CCSVI) in Patients With Multiple Sclerosis and Other Neurological Diseases
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Professor of Neurology, University at Buffalo
Other Study IDs: CDUS1
Record Dates: First submitted 2014-07-08; First posted 2014-12-04 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Clinically Isolated Syndrome (CIS); Multiple Sclerosis (MS); Other Neurological Disorders (OND); Healthy (HC)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Multiple Sclerosis: Patients diagnosed with Multiple Sclerosis (MS), identified in the CTEVD trial
- Clinically Isolated Syndrome: Patients diagnosed with Clinically Isolated Syndrome (CIS), identified in the CTEVD trial.
- Other Neurological Disorders: Patients diagnosed with Other Neurological Disorders (OND), identified in the CTEVD trial. ONDs fall into one of four categories: Neurodegenerative, Vascular, Autoimmune, and Neuromuscular; and the following disorders: Acute Disseminated Encephalomyelitis (ADEM); Antiphospholipid Antibody (syndrome; APLA); Atypical, short-lasting neurodegenerative disease; Autoimmune disease not otherwise specified (NOS); Cerebellum Syndrome; Charcot-Marie Tooth Disease; Chiari Malformation; Chronic Fatigue Syndrome; Central Nervous System Vasculitis; Demyelinating Disease; Epilepsy; Headaches; Idiopathic Chronic Neuropathy; Migraines; Mitochondrial Disease; Myelopathy; Neurofibromatosis; Neuropathy; Optic Neuritis; Parasthesia related to Transient Ischemic Attacks (TIA); Parkinson's Disease; Restless legs syndrome; Seizures; Spinal Cerebellum Disease; Spinal Disc Degeneration; Syringomyelia; and Vertigo
- Healthy Controls: Individuals who are healthy (i.e., free from neurological conditions; HC) , identified in the CTEVD trial.

SUMMARY:
This a retrospective, blinded trial in which collaborators in Italy will review the doppler findings from the Combined Transcranial and Extracranial Venous Doppler (CTEVD) trial in an attempt to measure reproducibility.

DETAILED DESCRIPTION:
This study will retrospectively investigate doppler images from the second phase of the CTEVD trial.

1. To determine the prevalence of CCSVI in patients with MS, compared with the prevalence observed in a control population consisting of Other Neurological Diseases (OND) patients and Healthy Controls (HC) by using blinded, controlled centralized ultrasound reading assessment of 5 Venous Haemodynamic (VH) CCSVI CCSVI Doppler UltraSound (CDUS) criteria.
2. To investigate whether prevalence of CCSVI is different between centralized and local CDUS reading of 5 VH CCSVI CDUS criteria.
3. To investigate the prevalence of CCSVI in patients with MS, compared with the prevalence observed in a control population consisting of OND patients and HC, when bidirectional flow in the intracranial veins and sinuses CDUS criterion is not considered as part of VH CCSVI CDUS criteria.
4. To determine whether prevalence of CCSVI in patients with MS, compared with the prevalence observed in a control population consisting of OND patients and HC differs when using CDUS velocity and flow parameters in the Internal Jugular Veins (IJVs) and Vertebral Veins (VVs).
5. To determine the reproducibility of VH criteria by using of centralized and local blinded, controlled CDUS reading assessment.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the CTEVD Phase 2 study
* Available CDUS exam
* Diagnosed with CIS, MS, OND, or being a HC
* Fulfilling inclusion criteria from the CTEVD study

Exclusion Criteria:

* Not having an available CDUS exam
* Diagnosed with Radiologically Isolated Syndrome (RIS) or Neuromyelitis Optic (NMO)
* Fulfilling exclusion criteria from the CTEVD study

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in this study will be those who had participated in the second phase of the Combined Transcranial/Extracranial Venous Deficiency (CTEVD) study.
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of MS (or CIS) and HC (or OND) who have 5 VH CCSVI CDUS criteria on doppler ultrasound | Baseline
  The prevalence (number) of MS/CIS vs. HC/OND who fulfill the 5 venous haemodynamic (VH) criteria on doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD, PhD, Principal Investigator — University at Buffalo